CLINICAL TRIAL: NCT00850551
Title: Early Intervention in Pulmonary Exacerbation in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Chris Goss, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35243-E/A
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: Early Intervention; Pulmonary Exacerbation; Cystic Fibrosis; Lung Function; Spirometry; Phillips Telemonitor; Home Spirometry; PiKo-6; Home Monitoring
MeSH Terms: conditions — Cystic Fibrosis | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Usual Care
  Interventions: Other: Early Intervention
- Intervention (Other): Twice weekly home spirometry and symptom assessment
  Interventions: Other: Early Intervention

INTERVENTIONS:
Other: Early Intervention — Twice a week home spirometry and symptom assessment
  Other Names: Piko-6; Philips Telemonitor

SUMMARY:
This study will be performed at the University of Washington. Forty subjects with Cystic Fibrosis will be enrolled, with 20 randomized into the usual care arm and 20 randomized into the intervention arm. All subjects will be enrolled for 6 months and have 3 study visits. One at baseline, midpoint, and final. The intervention arm subjects may have more study visits depending on their respiratory symptoms.

The intervention arm subjects will perform home spirometry twice a week with a PiKo-6 hand held spirometer. They will also have a home-based telemonitoring system connected to their phone line. They will be prompted twice a week to answer questions regarding their health via the telemonitor.

Subjects who are not able to utilize the home-based telemonitoring system will answer the questions regarding their health via the internet from their home computer.

If the subject's spirometry falls by greater than 10% from baseline or the CF respiratory symptoms change in 3 or more of the 8 respiratory symptoms captured by the telemonitor questionnaire, the subject will be called by the research staff and clinically evaluated by the study PIs within three days.

The usual care subjects will continue with their routine care at the University of Washington CF Clinic.

DETAILED DESCRIPTION:
The study design is a single center, randomized non-blinded controlled clinical trial comparing usual care to a program of early identification and treatment of pulmonary exacerbation in adults with CF. Forty subjects will be enrolled a at the University of Washington with 20 subjects randomized into the usual care arm, and 20 randomized into the intervention arm.

Usual care is defined as the regular quarterly CF visits with acute visits triggered by calls from the patient to the clinic. Neither home assessment of spirometry or standardized home symptom assessment are a component of usual care. Treatment of a pulmonary exacerbation will be based on a standard protocol employing a standard definition and treatment regimen. This study will employ current standardized CF pulmonary exacerbation orders used at the University of Washington. Usual care arm subjects will have 3 study visits at baseline, midpoint, and final, over a period of 6 months.

The early intervention protocol will employ twice a week assessment of home spirometry and CF respiratory symptoms; we will employ a home based monitoring system from Philips called the Philips Remote Patient Monitoring system (TeleStation). The home monitoring system is connected to the patient's phone line; this system is currently used in clinical practice in the care of patients with diabetes and heart failure.

Subjects who do not have a home phone line will answer the CF respiratory questions via the internet from their home computer.

The home spirometry will be done using a PiKo-6 hand held spirometer up to 84 spirometry values. If the subject's spirometry falls by greater than 10% from baseline or the CF respiratory symptoms change in 3 or more of the 8 respiratory symptoms captured in the questionnaire, the subject will be called by the research staff and clinically evaluated by the study PIs within three days. This evaluation will include a history and physical exam along with repeat spirometry at the clinic. The intervention arm subjects will have 3 study visits at baseline, midpoint, and final, over a period of 6 months. They may have additional study visits depending on their respiratory symptoms or exacerbations during the 6 month study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Confirmed diagnosis of cystic fibrosis
* Chronically colonization wtih Pseudomonas defined by positive sputum or lower airway cultures on 2 or more occasions in any 12 month period
* Ability to participate in an interview and administration of questionnaire lasting 60 minutes
* Clinically stable without IV antibiotic treatment for a pulmonary exacerbation in the prior 2 weeks
* Ability to perform spirometry
* Have a home telephone line or home computer with internet connection
* Written informed consent

Exclusion Criteria:

* Colonization with burkholderia cepacia complex
* Confirmed diagnosis of allergic bronchopulmonary aspergillosis as defined by the CFF guidance document
* Currently receiving antimicrobial therapy to treat non-tuberculous mycobacterium
* History of prior solid organ transplant
* Inability to speak and read the English language well enough to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of the use of home spirometry and home symptom assessment on the diagnosis of acute pulmonary exacerbation in adult patients with mild to moderate CF lung disease | 6 months

SECONDARY OUTCOMES:
Assess the impact of the use of home spirometry, home symptom assessment and a protocolized approach to treatment of acute pulmonary exacerbation compared to usual care. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Goss, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD